CLINICAL TRIAL: NCT02457416
Title: Take Away Food Allergy; Inducing Tolerance in Children Allergic to Peanut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Geir Håland, Consultant PhD/Post doc, Oslo University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/430
Record Dates: First submitted 2014-05-30; First posted 2015-05-29 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Food Hypersensitivity
Keywords: Peanut allergy; Oral immunotherapy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peanut oral immunotherapy (Active Comparator): Oral immunotherapy with peanut
  Interventions: Other: Peanut
- Controls (No Intervention): Avoid peanut exposure

INTERVENTIONS:
Other: Peanut — Treatment with peanut in increasing doses until a maintenance dose
  Arms: Peanut oral immunotherapy

SUMMARY:
The purpose of the study is to identify prognostic markers and possible success rate of tolerance induction to peanut allergens in children allergic to peanut.

DETAILED DESCRIPTION:
The study is an open randomized controlled study on oral immunotherapy including 60 children (40 on active treatment, 20 controls) with primary peanut allergy. The study has 4 phases: 1: inclusion/randomization including a double blind placebo controlled food Challenge 2: bi weekly up-dosing to maintenance dose after 48 weeks, 3: maintenance period of 3 years 4: 1 year follow up after end of treatment.

Clinical parameters as well as immunological (serological and cellular) will be recorded at inclusion, after 3 months of up-dosing, at end of up-dosing, after 1 and 3 years of maintenance treatment and after 3 and 12 year of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test or IgE to peanut
* Age 5-15 yrs
* Primary peanut allergy verified by objective symptoms to DBPCFC by a dose of 3 mg or more peanut potein

Exclusion Criteria:

* Non controlled asthma (by asthma control test, ACT)
* Allergy/intolerance to any other ingredients in the vehicle used for the peanut DBPCFC
* Current or previous allergen specific immunotherapy
* Cardiac disease with increased risk of serious anaphylaxis
* Severe atopic skin disease
* Diabetes mellitus
* Severe disease that interferes with adherence to study protocol

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2014-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with successfull tolerance induction to peanut | Data will be recorded for 5 years

SECONDARY OUTCOMES:
Clinical prognostic markers for successful tolerance induction to peanut | Data will be recorded for 5 years
  Clinical markers like severity of peanut allergy during double blind placebo controlled food challenge (DBPCFC), threshold level on DBPCFC, side effects during up dosing, maximum peanut dose reached, concomitant other atopic diseases will be assessed
Immunological prognostic markers for successful tolerance induction to peanut | Data will be recorded for 5 years
  Immunologic markers: Immunoglobulin E (IgE) to peanut and its components, total IgE, Immunoglobulin G4 to peanut and its components, Basophil activation test will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Geir Håland, MD PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Department of Paediatrics, Oslo, Norway

REFERENCES:
- [Derived] Reier-Nilsen T, Carlsen KCL, Michelsen MM, Drottning S, Carlsen KH, Zhang C, Borres MP, Haland G. Parent and child perception of quality of life in a randomized controlled peanut oral immunotherapy trial. Pediatr Allergy Immunol. 2019 Sep;30(6):638-645. doi: 10.1111/pai.13066. Epub 2019 Jul 25. PMID 31013372
- [Derived] Reier-Nilsen T, Michelsen MM, Lodrup Carlsen KC, Carlsen KH, Mowinckel P, Nygaard UC, Namork E, Borres MP, Haland G. Feasibility of desensitizing children highly allergic to peanut by high-dose oral immunotherapy. Allergy. 2019 Feb;74(2):337-348. doi: 10.1111/all.13604. Epub 2018 Oct 8. PMID 30225844